CLINICAL TRIAL: NCT06092450
Title: Deep Learning Radiomics Model for Predicting Post-cystectomy Outcome From Preoperative CT in Muscle Invasive Bladder Cancer
Brief Title: Deep Learning Radiomics Model for Predicting Post-cystectomy Outcome in Muscle Invasive Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Mingzhao Xiao, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: AI-BLCA; 2022-K508 (Other: The First Affiliated Hospital of Chongqing Medical University)
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
Keywords: Tomography, X-ray computed; Muscle-invasive bladder cancer; Radiomics; Deep Learning
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MIBC: patients with pathologically confirmed MIBC after radical cystectomy
  Interventions: Other: develop and validate a deep learning radiomics model based on preoperative enhanced CT image

INTERVENTIONS:
Other: develop and validate a deep learning radiomics model based on preoperative enhanced CT image — develop and validate a deep learning radiomics model based on preoperative enhanced CT to predict postoperative survival in MIBC

SUMMARY:
Muscle invasive bladder cancer (MIBC) has a poor prognosis even after radical cystectomy. Postoperative survival stratification based on radiomics and deep learning may be useful for treatment decisions to improve prognosis. This study was aimed to develop and validate a deep learning radiomics model based on preoperative enhanced CT to predict postoperative survival in MIBC.

ELIGIBILITY:
Inclusion Criteria:

* patients with pathologically confirmed MIBC after radical cystectomy;
* contrast-CT scan less than two weeks before surgery;
* complete CT image data and clinical data.

Exclusion Criteria:

* patients who received neoadjuvant therapy;
* non-urothelial carcinoma;
* poor quality of CT images;
* incomplete clinical and follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with pathologically confirmed MIBC who underwent radical cystectomy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival（OS） | up to 10 years
  the time from the date of surgery to death from any cause or the date of last contact (censored observation) at the date of data cut-off.
Recurrence free survival（RFS) | up to 10 years
  the time from the date of surgery to the date of first documented disease recurrence. Patients without recurrence at the time of analysis will be censored.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the current study are not publicly available due to the privacy of patients but are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Wei Z, Xv Y, Liu H, Li Y, Yin S, Xie Y, Chen Y, Lv F, Jiang Q, Li F, Xiao M. A CT-based deep learning model predicts overall survival in patients with muscle invasive bladder cancer after radical cystectomy: a multicenter retrospective cohort study. Int J Surg. 2024 May 1;110(5):2922-2932. doi: 10.1097/JS9.0000000000001194. PMID 38349205